CLINICAL TRIAL: NCT06817811
Title: Bioequivalence Study of Apixaban 5 mg Film-Coated Tablet Produced by PT Dexa Medica in Comparison With the Comparator Drug (Eliquis® 5 mg Film Coated Tablet, Bristol-Myers Squibb Company, Puerto Rico, Packed and Released By Bristol-Myers Squibb S.R.L., Italy, Imported by PT Pfizer Indonesia)
Brief Title: Bioequivalence Study of Apixaban 5 mg Film-Coated Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dexa Medica Group (Industry)
Collaborators: PT Equilab International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BE. 644/EQL/2020
Record Dates: First submitted 2025-02-05; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Health
MeSH Terms: interventions — apixaban; Product Packaging

STUDY DESIGN:
Intervention Model Description: This was a bioequivalence study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Apixaban 5 mg Film-Coated Tablet PT Dexa Medica (Experimental): Apixaban 5 mg Film-Coated Tablet (produced by PT Dexa Medica)
  Interventions: Drug: Apixaban 5 mg Film-Coated Tablet (produced by PT Dexa Medica)
- Reference Eliquis® 5 mg film-coated tablet, Bristol-Myers Squibb (Active Comparator): Eliquis® 5 mg film-coated tablet, Bristol-Myers Squibb Company, Puerto Rico, packed and released by Bristol-Myers Squibb S.r.l., Italy, imported by PT Pfizer Indonesia
  Interventions: Drug: Eliquis® 5 mg film-coated tablet (Bristol-Myers Squibb Company, Puerto Rico, packed and released by Bristol-Myers Squibb S.r.l., Italy, imported by PT Pfizer Indonesia)

INTERVENTIONS:
Drug: Apixaban 5 mg Film-Coated Tablet (produced by PT Dexa Medica) — One tablet of the test drug was given orally under fasting condition
  Arms: Test Apixaban 5 mg Film-Coated Tablet PT Dexa Medica
Drug: Eliquis® 5 mg film-coated tablet (Bristol-Myers Squibb Company, Puerto Rico, packed and released by Bristol-Myers Squibb S.r.l., Italy, imported by PT Pfizer Indonesia) — One tablet of the reference drug was given orally under fasting condition
  Arms: Reference Eliquis® 5 mg film-coated tablet, Bristol-Myers Squibb

SUMMARY:
This was an open-label, randomized, single-dose, two-period, two-sequence, cross-over study under fasting condition which included 24 healthy adult male and female subjects. The objective of this study was to find out whether the bioavailability of apixaban 5 mg film-coated tablet produced by PT Dexa Medica in comparison with the comparator drug (Eliquis® 5 mg filmcoated tablet, Bristol-Myers Squibb Company, Puerto Rico, packed and released by Bristol Myers Squibb S.r.l., Italy, imported by PT Pfizer Indonesia).

DETAILED DESCRIPTION:
The objective of this study was to find out whether the bioavailability of apixaban 5 mg film-coated tablet produced by PT Dexa Medica in comparison with the comparator drug (Eliquis® 5 mg filmcoated tablet, Bristol-Myers Squibb Company, Puerto Rico, packed and released by Bristol-Myers Squibb S.r.l., Italy, imported by PT Pfizer Indonesia). This was an open-label, randomized, single dose, two-period, two-sequence, cross-over study under fasting condition which included 24 healthy adult male and female subjects. The participating subjects were required to have an 8 hours overnight fast and in the next morning (first day of period) were given orally the test drug (apixaban 5 mg film-coated tablet produced by PT Dexa Medica) or the comparator drug (Eliquis® 5 mg Film Coated Tablet, Bristol-Myers Squibb Company, Puerto Rico, packed and released by Bristol-Myers Squibb S.r.l., Italy, imported by PT Pfizer Indonesia) with 200 mL of water. The subject's oral cavity was checked thoroughly to confirm complete medication and fluid consumption after dosing. Blood samples were drawn before taking the drug (control), and at 0.50, 1.00, 1.50, 2.00, 2.50, 3.00, 3.33, 3.67, 4.00, 4.50, 5.00, 6.00, 9.00, 12.00, 24.00, 36.00, and 48.00 hours after drug administration. These blood samples were used to investigate the pharmacokinetic parameters of apixaban following single dose administration. The plasma concentrations of apixaban were determined by using a validated ultra-performance liquid chromatography with tandem mass spectrometry detection (UPLC-MS/MS).

ELIGIBILITY:
Inclusion Criteria:

1. Able to participate, communicate well with the investigators and willing to provide written informed consent to participate in the study.
2. Healthy male and female subjects with absence of significant disease or clinically significant abnormal laboratory values on laboratory evaluation, medical history or physical examination during screening and could be considered healthy based on the evaluation.
3. Aged 18 - 55 years inclusive.
4. Preferably non-smokers or smoke less than 10 cigarettes per day.
5. Body mass index within 18 to 25 kg/m2.
6. Normal prothrombin time (PT) and normal partial thromboplastin time (aPTT)
7. Creatinine clearance > 50 mL/min
8. Vital signs (after 10 minutes rest) must be within the following ranges:

   * Systolic blood pressure: 100 - 129 mmHg
   * Diastolic blood pressure: 60 - 84 mmHg
   * Pulse rate: 60 - 90 bpm.

Exclusion Criteria:

1. History of allergy or hypersensitivity or contraindication to apixaban or factor Xa inhibitors or allied drug.
2. Pregnant or lactating female (urinary pregnancy test was applied to female subjects at screening and before taking the study drug).
3. Any major illness in the past 90 days or clinically significant ongoing chronic medical illness.
4. Presence of any clinically significant abnormal values during screening e.g. significant abnormality of liver function test (AST, ALT, alkaline phosphatase, total bilirubin, direct bilirubin ≥ 1.5 ULN), renal function test (serum creatinine concentration > 1.4 mg/dL and ureum ≥ 1.5 ULN), etc.
5. Positive Hepatitis B surface antigen (HBsAg), anti-HCV, or anti-HIV.
6. Clinically significant hematology abnormalities.
7. Positive result for COVID-19 antigen rapid test.
8. Clinically significant electrocardiogram (ECG) abnormalities.
9. Any surgical or medical condition (present or history) which might significantly alter the absorption, distribution, metabolism or excretion of the study drug, e.g. gastrointestinal disease including gastric or duodenal ulcers or history of gastric surgery.
10. Past history of anaphylaxis or angioedema.
11. History of drug or alcohol abuse within 12 months prior to screening for this study.
12. Participation in any clinical trial within the past 90 days calculated from the last visit until this study's first dosing day.
13. History of any bleeding or coagulative disorders.
14. History of significant head injury within the last two years.
15. Presence of difficulty in accessibility of veins in left or right arm.
16. A donation or significant blood loss within 90 days before this study's first dosing day.
17. Intake of any prescription, (especially apixaban, other anticoagulants, azole antimycotics), non-prescription drug, (including hormonal contraception), food supplements or herbal medicines within 21 days of this study's first dosing day

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2021-04-24 (Actual); Study Completion 2021-06-03 (Actual)

PRIMARY OUTCOMES:
AUC(0-t) | 48 hours
  Area under the plasma concentration-time curve to the last observer quantifiable concentration at time t
Cmax | 48 hours
  Maximum plasma concentration

SECONDARY OUTCOMES:
AUC(0-inf) | 48 hours
  Area under the plasma concentration-time curve extrapolated to infinitive time
T1/2 | 48 hours
  Plasma half-life
Tmax | 48 hours
  Time taken to reach maximum observed plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Danang A Yunaidi, Principal Investigator — PT Equilab International
Locations (1):
- PT Equilab International, Jakarta, Indonesia